CLINICAL TRIAL: NCT03312569
Title: A Multi-Center Prospective Comparison of Intracorporeal and Extracorporeal Anastomoses for Minimally Invasive Right Colectomy
Brief Title: Robotic-assisted and Laparoscopic Right Colectomy Study - Intracorporeal vs. Extracorporeal Anastomoses
Acronym: ANCOR
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVRC-002
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Benign Right Colon Disease; Malignant Right Colon Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Intracorporeal Anastomosis: Participants will undergo either robotic-assisted or laparoscopic surgery with an intracorporeal anastomosis due to begin or malignant Right Colon Disease.
  Interventions: Procedure: Right Colectomy with Intracorporeal Anastomosis
- Extracorporeal Anastomosis: Participants will undergo either robotic-assisted or laparoscopic surgery with an extracorporeal anastomosis due to begin or malignant Right Colon Disease.
  Interventions: Procedure: Right Colectomy with Extracorporeal Anastomosis

INTERVENTIONS:
Procedure: Right Colectomy with Intracorporeal Anastomosis — With the patient under general anesthesia, pneumoperitoneum is achieved by a method of choice of the operating surgeon. Port Placement is completed as per the standard of care. Dissection is performed and the ileocolic vessels are identified. The right mesocolon is mobilized and the ileal mesentery is divided. The transverse colon and ileum are then divided with the stapler. Next, attention is turned to constructing the anastomosis. For this purpose, the terminal ileum and the transverse colon stump are brought together. A colotomy and ileostomy is created to form a common channel. The common enterotomy is then closed as per the surgeon's standard of care. The specimen is extracted through an off-midline incision (muscle splitting transverse incision, Pfannenstiel).
  Groups: Intracorporeal Anastomosis
Procedure: Right Colectomy with Extracorporeal Anastomosis — With the patient under general anesthesia, pneumoperitoneum is achieved by a method of choice of the operating surgeon. Port Placement is completed as per the standard of care. Dissection is performed and the ileocolic vessels are identified. Intracorporeal devascularization may be performed at the surgeon's discretion. The gastrocolic ligament is taken down and the hepatic flexure is mobilized. After complete mobilization of the right colon, the midline incision is extended to serve as the extraction site. The specimen is delivered through the midline extraction incision and the anastomosis is conducted in a standard open technique. The two cut ends of the bowels are aligned for extracorporeal anastomosis.
  Groups: Extracorporeal Anastomosis

SUMMARY:
To compare intracorporeal and extracorporeal anastomoses for robotic-assisted and laparoscopic right colectomies

DETAILED DESCRIPTION:
This is a prospective multicenter observational study to evaluate outcomes of intracorporeal and extracorporeal anastomoses for robotic-assisted and laparoscopic right colectomies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject undergoing either laparoscopic or robotic-assisted right colectomy for benign or malignant right colon disease
* Subject undergoing intracorporeal or extracorporeal anastomosis proximal to mid-transverse colon

Exclusion Criteria:

* Subject is contraindicated for general anesthesia or surgery
* Emergent Case
* Subject has perforated, obstructing or locally invasive neoplasm (T4b)
* Subject with inflammatory bowel disease
* Subject with prior incisional hernia repair
* Planned right colectomy along with major concomitant procedures (e.g. hepatectomies, other intestinal resections).
* Metastatic disease with life expectancy of less than 1 year
* Pregnant or suspect pregnancy
* Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
* Subject belonging to other vulnerable population, e.g, prisoner or ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject undergoing either laparoscopic or robotic-assisted right colectomy for benign or malignant right colon disease
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Incidence of incisional hernia at one year after index procedure. | 1 year
  The primary endpoint of the study is the incidence of incisional hernia for intracorporeal and extracorporeal anastomoses within one year after the right colectomy procedure. Incidence of incisional hernia either patient self-reported or clinical diagnosis will be assessed at one year after the right colectomy procedure.

SECONDARY OUTCOMES:
Time to first flatus after index procedure | up to 1 week after index procedure
  The secondary endpoint of the study is time to first flatus for intracorporeal and extracorporeal anastomoses after the right colectomy procedure. Time to first flatus is defined as days from a right colectomy procedure to first occurrence of flatus during subject's post-operative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Mehendale, Study Director — Intuitive Surgical Inc
Locations (4):
- United States (4):
  - University of California, Irvine, California
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Washington University at St. Louis, St Louis, Missouri
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cleary RK, Silviera M, Reidy TJ, McCormick J, Johnson CS, Sylla P, Cannon J, Lujan H, Kassir A, Landmann RG, Gaertner W, Lee E, Bastawrous AL, Bardakcioglu O, Pandey S, Attaluri V, Bernstein M, Obias V, Pigazzi A. Extraction site hernia and short-term outcomes following intracorporeal versus extracorporeal anastomosis for robotic and laparoscopic right colectomy: a multi-center prospective trial. Surg Endosc. 2026 Jan;40(1):502-511. doi: 10.1007/s00464-025-12327-7. Epub 2025 Oct 27. PMID 41145697